CLINICAL TRIAL: NCT00714506
Title: Effects of a Weight Reduction and Lifestyle Program in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Anne B. Newman, Professor of Epidemiology, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: PRO07040024
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Functional Disability; Obesity; Physical Inactivity
Keywords: obesity; physical activity; older adults; functional disability
MeSH Terms: conditions — Obesity; Sedentary Behavior; Motor Activity | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): lifestyle weight reduction - low fat eating, low calorie and physical activity
  Interventions: Behavioral: Diet and physical activity
- Control (Active Comparator): physical activity plus successful aging health education
  Interventions: Other: Physical activity control

INTERVENTIONS:
Behavioral: Diet and physical activity — lifestyle weight reduction - low fat eating, low calorie and physical activity
  Arms: Intervention
Other: Physical activity control — physical activity plus successful aging health education
  Arms: Control

SUMMARY:
This research study will assess the effects of two different programs on weight, body composition, mobility and improved health. Measures of health will include functional abilities, and physical performance. The 2 programs being tested will be provided the same physical activity program which will include aerobic activity and resistance (weight) training. The intervention study will last up to 1 year with follow-up at 6 months and yearly phone calls thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and older
* BMI 28 to 39.9
* Sedentary lifestyle defined by formal exercise less than 3 times per week for a total of less than 90 minutes.
* Self report of ability to walk ¼ mile (2-3 blocks)
* Ability to complete the 400 meter walk without a cane or walker in less than 15 minutes
* Successful completion of the behavioral run-in phase which includes an activity log and a food diary
* Willingness to be randomized to either intervention group
* Willingness to attend meetings and physical activity sessions in McKeesport

Exclusion Criteria:

* Diabetes requiring insulin, history of diabetic coma, or diabetes out of control defined as fasting blood sugar greater than 300
* Severe hypertension, e.g. SBP> 180, DBP > 100
* Failure to provide informed consent
* Nursing home resident or resident in a facility where they have no control over food choices
* Significant cognitive impairment, defined as a known diagnosis of dementia or a 3MSE Cognitive Function score < 80
* Major psychiatric disorder
* Unable to communicate because of severe hearing loss or speech disorder
* Severe visual impairment
* Celiac sprue or other malabsorption syndromes
* Consume more than 5 alcoholic drinks per day, or more than 15 drinks per week
* Progressive, degenerative neurological disease
* Severe rheumatologic or orthopedic diseases
* Stroke, hip, or knee replacement, or spinal surgery within the past 4 months or planned in the next 4 months
* Receiving physical therapy for gait, balance, or lower extremity training
* Terminal illness with life expectancy of less than 12 months
* Currently being treated with chemotherapy or radiation for breast, cervical, colon, prostate, rectal, uterine, thyroid, or oral cancer. Participant with other types of cancers, with the exception of basal and squamous cancer are ineligible
* Severe pulmonary disease (i.e., lung disease requiring supplemental oxygen or oral steroid medication) or pulmonary embolism or deep vein thrombosis within the past 6 months
* Severe cardiac disease (i.e., congestive heart failure (NYHA Class III or IV); untreated aortic stenosis; a history of cardiac arrest, the use of a cardiac defibrillator or uncontrolled angina)
* Myocardial infarction, CABG, or valve replacement in the past 6 months
* Serious conduction disorder (3rd degree heart block), uncontrolled arrhythmia, or new Q waves or ST- segment depressions (> 3mm) on ECG
* Other significant co-morbid disease that the study medical officer deems severe enough to impair ability to participate in exercise based intervention
* Severe kidney disease that requires dialysis
* Develops chest pain or severe shortness of breath during 400 m walk test
* Member of household is already enrolled
* Participation in another intervention trial: participation in an observational study is permitted
* People who have lost more than 10 pounds in the past 4 months, or are on any drugs for the treatment of obesity
* Lives outside of the study site area or is planning to move in the next year
* Must be able to attend at least 6 of the first 8 weekly sessions.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
time to walk 400 m | at 6 mo intervals

SECONDARY OUTCOMES:
weight loss | 6 month intervals

CONTACTS AND LOCATIONS:
Overall Officials: Anne B Newman, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- McKeesport Hospital - Kelly Building, McKeesport, Pennsylvania, United States

REFERENCES:
- [Derived] Farsijani S, Cauley JA, Santanasto AJ, Glynn NW, Boudreau RM, Newman AB. Transition to a More even Distribution of Daily Protein intake Is Associated with Enhanced Fat Loss during a Hypocaloric and Physical Activity Intervention in Obese Older Adults. J Nutr Health Aging. 2020;24(2):210-217. doi: 10.1007/s12603-020-1313-8. PMID 32003413
- [Derived] Santanasto AJ, Newman AB, Strotmeyer ES, Boudreau RM, Goodpaster BH, Glynn NW. Effects of Changes in Regional Body Composition on Physical Function in Older Adults: A Pilot Randomized Controlled Trial. J Nutr Health Aging. 2015 Nov;19(9):913-21. doi: 10.1007/s12603-015-0523-y. PMID 26482693